CLINICAL TRIAL: NCT01752777
Title: Behavioral Intervention to Enhance HIV Test/Treat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Seth Kalichman, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H11-159
Record Dates: First submitted 2012-12-16; First posted 2012-12-19 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS, HIV infectiousness, Medication adherence, Sexual risks reduction
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infectiousness Risk Reduction (Experimental): Behavioral counseling conducted in one office session followed by 4 cell-phone-based sessions. Counseling is based on models of behavioral self-management and cognitive decision making with the primary aim to increase antiretroviral adherence, engagement in HIV care, and reduction of sexual risk behaviors for HIV transmission.
  Interventions: Behavioral: Infectiousness Risk Reduction
- General Health Improvement (Sham Comparator): Participants in this condition receive education conducted in one office session followed by 4 cell-phone-based sessions. The education sessions focus on raising awareness of health services and health improvement strategies.
  Interventions: Behavioral: General Health Improvement

INTERVENTIONS:
Behavioral: Infectiousness Risk Reduction — Behavioral counseling conducted in one office session followed by 4 cell-phone-based sessions. Counseling is based on models of behavioral self-management and cognitive decision making with the primary aim to increase antiretroviral adherence, engagement in HIV care, and reduction of sexual risk behaviors for HIV transmission.
  Arms: Infectiousness Risk Reduction
Behavioral: General Health Improvement — Educational counseling to help link participants to social serves and health related strategies.
  Arms: General Health Improvement

SUMMARY:
Prevention strategies that aim to test and treat people for HIV infection are undermined by HIV treatment non-adherence and sexually transmitted co-infections (STI). The proposed study will test a theory-based behavioral intervention to reduce HIV infectiousness by simultaneously improving HIV treatment adherence and reducing sexually transmitted co-infections in people living with HIV-AIDS who use alcohol and other drugs. The intervention is delivered in a single office-based counseling session followed by 4 cell phone delivered counseling sessions in a model that will be ready for immediate dissemination to case management and clinical services for people living with HIV/AIDS in resource constrained settings.

DETAILED DESCRIPTION:
Prevention strategies that aim to test and treat people for HIV infection are undermined by HIV treatment non-adherence and sexually transmitted co-infections (STI). Scalable interventions are urgently needed to sustain low infectiousness by improving HIV treatment adherence and reducing risks for transmitting HIV. This application proposes to test a theory-based behavioral intervention to simultaneously improve HIV treatment adherence and reduce HIV transmission risk behaviors in people living with HIV/AIDS who use alcohol and other drugs. Grounded in Conflict Theory of Decision Making, the intervention will be delivered in a mixed format, with one office-based counseling session followed by four cell phone delivered counseling sessions. The intervention will be conducted in Atlanta and surrounding impoverished areas. Men (n = 250) and women (n = 250) receiving HIV treatment will be recruited from AIDS services and infectious disease clinics. Following informed consent and baseline assessments, participants will be randomly assigned to either an (a) integrated HIV treatment adherence - risk reduction intervention or (b) a time-matched non-contaminating attention control condition. Participants will be followed for 12-months using office-based computerized interviews, unannounced pill counts, and medical chart abstraction. The study will test the hypothesis that a unified, integrated theory-based HIV treatment and risk reduction intervention will reduce HIV transmission risk behaviors, improve HIV treatment adherence, reduce viral load and prevent new STI. The study will also examine the influence of theoretical constructs and structural barriers on intervention outcomes. Factors that predict relapse to non-adherence and risk behaviors in relation to changes in viral load and STI over the 12-month follow-up period will also be a focal point of the study. The intervention under investigation will be among the first to simultaneously address treatment adherence and risk behavior in an integrated model for substance using HIV positive men and women. If shown effective, the intervention model will be ready for immediate dissemination to community and clinical services for people living with HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* HIV positive
* Sexually active in the previous Month
* Active substance use

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
HIV RNA Viral Load | 12 month
  HIV RNA viral load determined by blood plasma PCR

SECONDARY OUTCOMES:
Sexual Transmission Risk Behaviors | 3 month
  Sexual behaviors that create risks for HIV transmission and protective actions against transmission risks

CONTACTS AND LOCATIONS:
Locations (1):
- Southeast HIV/AIDS Research and Evaluation Project, Atlanta, Georgia, United States